CLINICAL TRIAL: NCT05408312
Title: Phase I Clinical Trial of Safety, Tolerance and Immunogenicity of GEN2-Recombinant COVID-19 Vaccine (CHO Cells) in Healthy People Aged 18 and Above
Brief Title: Phase I Clinical Trial of GEN2-Recombinant COVID-19 Vaccine (CHO Cells) in Healthy People Aged 18 and Above
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Vaccine and Serum Institute, China (Industry)
Collaborators: Lanzhou Institute of Biological Products Co., Ltd (Industry); Beijing Institute of Biological Products Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CXSL2200156-Ⅰ
Record Dates: First submitted 2022-06-05; First posted 2022-06-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group 1 (Experimental)
  Interventions: Biological: Experimental Vaccine 1
- Experimental group 2 (Experimental)
  Interventions: Biological: Experimental Vaccine 2
- Experimental group 3 (Experimental)
  Interventions: Biological: Experimental Vaccine 3
- placebo group (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Experimental Vaccine 1 — Intramuscular injection of low-dose Recombinant SARS-CoV-2 Vaccine (CHO cells，NVSI-06-08) in the deltoid muscle of the upper arm
  Arms: Experimental group 1
Biological: Experimental Vaccine 2 — Intramuscular injection of low-dose Recombinant SARS-CoV-2 Vaccine (CHO cells，NVSI-06-08) in the deltoid muscle of the upper arm
  Arms: Experimental group 2
Biological: Experimental Vaccine 3 — Intramuscular injection of low-dose Recombinant SARS-CoV-2 Vaccine (CHO cells，NVSI-06-08) in the deltoid muscle of the upper arm
  Arms: Experimental group 3
Biological: placebo — Intramuscular injection of low-dose Recombinant placebo in the deltoid muscle of the upper arm
  Arms: placebo group

SUMMARY:
phase I study will evaluate the safety and tolerability of GEN2-Recombinant COVID-19 Vaccine (CHO cells) in healthy people aged 18 years and older.

A total of 234 subjects were enrolled, of which 126 were enrolled in the 18-59-year-old group, and were randomly assigned to receive experimental vaccine 1, experimental vaccine 2, experimental vaccine 3 and placebo in a ratio of 2:2:2:1; 60- A total of 54 people were enrolled in the 69-year-old and ≥70-year-old groups, and were randomly assigned to receive the experimental vaccine 1 and placebo according to the ratio of 2:1.

ELIGIBILITY:
Inclusion Criteria:

* Age range: healthy people aged 18 and above, who can provide legal identification;
* No history of t SARS-CoV-2 vaccination;
* Able to provide a negative nucleic acid test certificate for the new coronavirus within 48 hours;
* Have the ability to understand (if illiterate, a fair witness is required to accompany the informed consent) research procedures, have informed consent, voluntarily sign the informed consent form, and be able to comply with the requirements of the clinical research protocol；
* Inquire about medical history and physical examination, and the investigator judges that the health status is good;
* Females of childbearing age (menarche to menopause) were not pregnant (negative urine pregnancy test) at enrollment, were not breastfeeding, and had no reproductive plans within the first 6 months after enrollment and took effective contraceptive measures; 2 weeks prior to enrollment have taken effective contraceptive measures;
* Able and willing to complete the entire prescribed study plan throughout the study follow-up period.

Exclusion Criteria:

First-dose exclusion criteria：

* Confirmed cases, suspected cases, asymptomatic infections, or close contacts of the above-mentioned groups of SARS-CoV-2 infection (check "China Disease Prevention and Control Information System");
* Axillary body temperature ≥37.3℃ before vaccination;
* Positive test for novel coronavirus antibody (IgG+IgM);
* Have a history of SARS virus infection (self-report, on-site inquiry);
* Fever (axillary temperature ≥37.3℃), dry cough, fatigue, nasal congestion, runny nose, sore throat, myalgia, diarrhea, shortness of breath, and dyspnea within 14 days before vaccination;
* The test results of blood biochemistry, blood routine, urine routine and coagulation function-related indexes before vaccination are abnormal, which are beyond the reference value range and have clinically significant abnormalities;
* Severe allergic reactions (such as acute allergic reactions, urticaria, skin eczema, dyspnea, angioedema or abdominal pain) have occurred in the past;
* Allergy to any component of the study vaccine (such as: aluminum, histidine, etc.);
* Patients with convulsions, epilepsy, encephalopathy or other progressive neurological diseases (such as transverse myelitis, Guillain-Barre syndrome, demyelinating diseases, etc.), long-term history of alcohol and drug abuse, history of thyroidectomy, infectious diseases, mental illness medical or family history;
* Known or suspected diseases include: severe respiratory disease, severe liver and kidney disease, severe cardiovascular disease, uncontrolled hypertension (systolic blood pressure ≥140mmHg, diastolic blood pressure ≥90mmHg), diabetic complications, malignant tumors, Various acute diseases, acute exacerbations of chronic diseases or severe chronic diseases;
* Have been diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;
* Thrombocytopenia, history of abnormal coagulation function (such as coagulation factor deficiency, coagulation disease);
* Asplenia or splenectomy, functional asplenia caused by any circumstance;
* Are receiving anti-TB (tuberculosis) treatment;
* Received immune enhancement or inhibitor therapy within 3 months (continuous oral or infusion for more than 14 days);
* Received live attenuated vaccine within 28 days before vaccination, and received other vaccines within 14 days before vaccination;
* Received blood products within 3 months before vaccination;
* Received other study drugs within 6 months before vaccination;
* Planning to move before the end of the study or to be away from the local area for an extended period of time during a scheduled study visit;
* The investigator judges other circumstances that are not suitable to participate in this clinical trial.

Exclusion criteria for second and third doses：

* Positive urine pregnancy test;
* Patients with abnormal conditions such as high fever (axillary temperature ≥39.0℃) for three days, convulsions, severe allergic reactions or any adverse reactions of the --Nervous system after the previous dose of vaccination;
* Serious adverse reactions that are causally related to the previous dose of vaccination;
* For those newly discovered or newly discovered after the previous dose of vaccine that do not meet the first-dose inclusion criteria or meet the first-dose exclusion criteria, the investigator will determine whether to continue participating in the study;
* Other reasons for exclusion considered by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2022-06-18 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
The incidence rate of any adverse reactions/events | within 30 minutes after vaccination
The incidence severity of any adverse reactions/events | within 30 minutes after vaccination
the incidence of abnormal blood biochemistry, blood routine, blood coagulation function and urine routine | on the 4th day after each dose of vaccination
The incidence rate of solicited adverse reactions/events | within 0-7 days after vaccination
The incidence severity of solicited adverse reactions/events | within 0-7 days after vaccination
The incidence rate of solicited adverse reactions/events | within 8-30 days after vaccination
The incidence severity of solicited adverse reactions/events | within 8-30 days after vaccination
Incidence of adverse events leading to withdrawal | within 8-30 days after vaccination
Severity of adverse events leading to withdrawal | within 8-30 days after vaccination
The incidence of SAE observed | up to 12 months after full course of immunization
The incidence of AESI observed | up to 12 months after full course of immunization
Neutralizing antibody level against SARS-CoV-2 GMT | Day 15th, 30th, 90th, 180th, 270th, 360th after full course of immunization
Neutralizing antibody level against SARS-CoV-2 IgG antibody GMC | Day 15th, 30th, 90th, 180th, 270th, 360th after full course of immunization
Neutralizing antibody level against SARS-CoV-2 positive rate | Day 15th, 30th, 90th, 180th, 270th, 360th after full course of immunization
Neutralizing antibody level against SARS-CoV-2 Positive conversion rate | Day 15th, 30th, 90th, 180th, 270th, 360th after full course of immunization

SECONDARY OUTCOMES:
GMT of GEN2-Recombinant COVID-19 Vaccine (CHO cells, NVSI-06-08) against VOC in healthy people aged 18 and above | after the full course of immunization
Cellular immune response level of subjects aged 18-59 | Before the first vaccination ， 15 days after the full course of immunization

CONTACTS AND LOCATIONS:
Locations (1):
- Ning ling Center for Disease Control and Prevention, Shangqiu, Henan, China

IPD SHARING:
Plan to Share IPD: No